CLINICAL TRIAL: NCT00068393
Title: Phase II Trial of Doxorubicin and Gemcitabine in Metastatic Renal Cell Carcinoma With Sarcomatoid Features
Brief Title: Doxorubicin and Gemcitabine in Treating Patients With Locally Recurrent or Metastatic Unresectable Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000322258; E8802 (Other: Eastern Cooperative Oncology Group (ECOG)); U10CA021115 (NIH)
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Results first posted 2013-01-04 (Estimated); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Metastatic Renal Cell Carcinoma; Renal Cell Carcinoma With Sarcomatoid Features
Keywords: Sarcomatoid; Gemcitabine; Doxorubicin; Renal cell cancer; Kidney cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Doxorubicin; Gemcitabine; Granulocyte Colony-Stimulating Factor; Filgrastim; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Doxorubicin/Gemcitabine (Experimental): Doxorubicin was given at 50 mg/m² by IV slow push, followed by gemcitabine 1500 mg/m² IV infusion over 30 minutes on day 1. Patients will receive G-CSF at a subcutaneous dose of 5mcg/kg/day on days 2 or 3 to 10 or neulasta at a dose of 6mg on day 2. Growth factor must be administered as close as possible to 24 hours after the completion of chemotherapy. It is recommended that neulasta be administered only on day 2 due to its prolonged half-life. Cycles were repeated every 2 weeks.
  Interventions: Drug: Doxorubicin; Drug: Gemcitabine; Drug: G-CSF (granulocyte-colony stimulating factor); Drug: Neulasta

INTERVENTIONS:
Drug: Doxorubicin — Doxorubicin: 50 mg/m² IV slow push followed by gemcitabine 1500 mg/m² IV infusion over 30 minutes on day 1. Cycles repeat every 2 weeks.
  Other Names: Adriamycin; Rubex
Drug: Gemcitabine — Doxorubicin: 50 mg/m² IV slow push followed by gemcitabine 1500 mg/m² IV infusion over 30 minutes on day 1. Cycles repeat every 2 weeks.
Drug: G-CSF (granulocyte-colony stimulating factor) — Patients will receive G-CSF at a subcutaneous dose of 5mcg/kg/day on days 2 or 3 to 10 or neulasta at a dose of 6mg on day 2. Growth factor must be administered as close as possible to 24 hours after the completion of chemotherapy. It is recommended that neulasta be administered only on day 2 due to its prolonged half-life.
  Other Names: Neupogen; Filgrastim
Drug: Neulasta — Patients will receive G-CSF at a subcutaneous dose of 5mcg/kg/day on days 2 or 3 to 10 or neulasta at a dose of 6mg on day 2. Growth factor must be administered as close as possible to 24 hours after the completion of chemotherapy. It is recommended that neulasta be administered only on day 2 due to its prolonged half-life.
  Other Names: pegfilgrastim

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin and gemcitabine, use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving doxorubicin together with gemcitabine works in treating patients with locally recurrent or metastatic unresectable renal cell carcinoma (kidney cancer).

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of patients with locally recurrent or metastatic unresectable renal cell cancer with sarcomatoid features treated with doxorubicin and gemcitabine.
* Determine the progression-free survival and overall survival of patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive doxorubicin intravenously (IV) and gemcitabine IV over 30 minutes on day 1. Patients also receive filgrastim (G-CSF) subcutaneously (SC) on days 2- or 3-10 or pegfilgrastim SC on day 2. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.

After 6 courses, patients undergo a MUGA scan. Patients with a stable* left ventricular ejection fraction (LVEF) continue therapy as above. Patients who reach a total doxorubicin dose of 450 mg/m^2 and are found to have unstable cardiac function or who have an abnormal LVEF continue therapy with gemcitabine alone.

NOTE: *Stable cardiac function is defined as no decrease more than 15% of LVEF in absolute number and LVEF at least 35% in total function by MUGA.

Patients are followed every 3 months for 2 years and then every 6 months for 1 year.

ACTUAL ACCRUAL: A total of 39 patients were accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA:

* Histologically confirmed renal cell carcinoma

  * Features must be of sarcomatoid histology
  * Locally recurrent or metastatic disease not amenable to resection
* Measurable disease
* Must have a prior nephrectomy provided all other eligibility criteria are met, and adequately recovered from any recent surgery
* At least 4 weeks since prior radiotherapy and recovered
* ECOG performance status of 0-1
* WBC greater than 3,000/mm^3 or absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3
* Bilirubin less than 1.5 mg/dL
* Aspartate aminotransferase (AST) less than 2 times upper limit of normal
* Creatinine no greater than 2.0 mg/dL
* LVEF at least lower limit of normal by MUGA
* Negative pregnancy test
* Fertile patients must use effective contraception
* Other prior malignancy allowed provided patient was curatively treated and has been disease free from that cancer
* Age of 18 and over
* Diagnostic material from the kidney or metastatic site biopsy available for central pathologic review

EXCLUSION CRITERIA:

* Prior treatment for advanced disease
* Previously irradiated lesions as the sole site of disease for patients with prior radiation therapy
* Concurrent local radiotherapy for pain control or for life-threatening situations
* Myocardial infarction within the past year
* Congestive heart failure within the past year
* Significant ischemic or valvular heart disease within the past year
* Prior or concurrent brain metastases
* Concurrent serious medical illness that would preclude study treatment
* Active infection that would preclude study treatment
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2004-02-24 (Actual); Primary Completion 2009-06 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naomi S. Balzer-Haas, MD, Study Chair — Fox Chase Cancer Center
Locations (92):
- United States (92):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Hematology/Oncology of the North Shore at Gross Point Medical Center, Skokie, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - William N. Wishard Memorial Hospital, Indianapolis, Indiana
  - Howard Community Hospital at Howard Regional Health System, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Miller-Dwan Medical Center, Duluth, Minnesota
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Hematology-Oncology Associates of Central New York, Syracuse, New York
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - St. Rita's Medical Center, Lima, Ohio
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Central Pennsylvania Hematology and Medical Oncology Associates, PC, Lemoyne, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Community Comprehensive Cancer Center at Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Medical Consultants, Limited, Milwaukee, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Haas N, Manola J, Pins M, et al.: ECOG 8802: phase II trial of doxorubicin (Dox) and gemcitabine (Gem) in metastatic renal cell carcinoma (RCC) with sarcomatoid features. [Abstract] J Clin Oncol 27 (Suppl 15): A-5038, 2009.
- [Result] Haas NB, Lin X, Manola J, Pins M, Liu G, McDermott D, Nanus D, Heath E, Wilding G, Dutcher J. A phase II trial of doxorubicin and gemcitabine in renal cell carcinoma with sarcomatoid features: ECOG 8802. Med Oncol. 2012 Jun;29(2):761-7. doi: 10.1007/s12032-011-9829-8. Epub 2011 Feb 6. PMID 21298497

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on December 9, 2003, accrued its first patient on February 24, 2004, and was closed to accrual on April 19, 2007. A total of 39 patients were registered to the study.
Groups:
- Doxorubicin/Gemcitabine: Doxorubicin was given at 50 mg/m² by IV slow push, followed by gemcitabine 1500 mg/m² IV infusion over 30 minutes on day 1. Patients will receive G-CSF at a subcutaneous dose of 5mcg/kg/day on days 2 or 3 to 10 or neulasta at a dose of 6mg on day 2. Growth factor must be administered as close as possible to 24 hours after the completion of chemotherapy. It is recommended that neulasta be administered only on day 2 due to its prolonged half-life. Cycles were repeated every 2 weeks.
  Only eligible and treated patients are included in the analysis.
Period: Overall Study
Arm/Group | Doxorubicin/Gemcitabine
Started | 39
Eligible and Treated | 38
Completed | 29
Not Completed | 10
Not completed — Adverse Event | 2
Not completed — Death | 3
Not completed — Withdrawal by Subject | 3
Not completed — Alternative treatment | 1
Not completed — Quality of life worsening | 1

BASELINE CHARACTERISTICS:
Arm/Group | Doxorubicin/Gemcitabine
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 59 [36 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 30
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Response Rate by Solid Tumor Response Criteria (RECIST)
Description: Per RECIST criteria, Complete response (CR)= disappearance of all target and nontarget lesions Partial response (PR)= >=30% decrease in the sum of the longest diameters of target lesions from baseline, and persistence of one or more non-target lesion(s) and/or the maintenance of tumor marker level above the normal limits. Objective response = CR + PR
Time Frame: Every 8 weeks during treatment; then every 3 months if <2 years from study entry; then every 6 months if 2-3 years from study entry
Population: Only eligible and treated patients are included in this analysis.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Doxorubicin/Gemcitabine
Number analyzed (Participants) | 38
Percentage of Participants | 16 [7 to 29]

2. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from study entry until death from any cause.
Time Frame: Every 2 weeks during treatment; then every 3 months if <2 years from study entry; then every 6 months if 2-3 years from study entry
Population: Only eligible and treated patients are included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Doxorubicin/Gemcitabine
Number analyzed (Participants) | 38
Months | 8.8 [6.1 to 11.1]

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as time from study entry until disease progression or death from any cause, whichever occurs first. Progression is defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of one or more new lesion(s) or unequivocal progression of existing nontarget lesions.
Time Frame: as for outcome 1
Population: Only eligible and treated patients are included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Doxorubicin/Gemcitabine
Number analyzed (Participants) | 38
Months | 3.5 [2.2 to 5.2]

ADVERSE EVENTS:
Time Frame: Assessed every 2 weeks while on treatment and for 30 days after the end of treatment.
Arm/Group | Doxorubicin/Gemcitabine
Serious Adverse Events (participants affected / at risk) | 15/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Doxorubicin/Gemcitabine (N=38)
Anemia (Blood and lymphatic system disorders) | 5
Leukopenia (Investigations) | 4
Neutropenia (Investigations) | 7
Thrombocytopenia (Investigations) | 1
Atrial fibrillation (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Fatigue (General disorders) | 3
Death - multiorgan failure (General disorders) | 1
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Infection w/ Gr0-2 neutropenia, lung (Infections and infestations) | 1
Infection w/ unknown ANC peristomal (Infections and infestations) | 1
Infection w/ unknown ANC upper airway NOS (Infections and infestations) | 1
Infection w/ unknown ANC urinary tract NOS (Infections and infestations) | 1
Chest wall, pain (Musculoskeletal and connective tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Doxorubicin/Gemcitabine (N=38)
Anemia (Blood and lymphatic system disorders) | 32
Leukopenia (Investigations) | 7
Lymphopenia (Investigations) | 2
Neutropenia (Investigations) | 3
Thrombocytopenia (Investigations) | 7
Left ventricular systolic dysfunction (Cardiac disorders) | 2
Fatigue (General disorders) | 27
Fever w/o neutropenia (General disorders) | 4
Weight loss (Investigations) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 22
Nail changes (Skin and subcutaneous tissue disorders) | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 15
Constipation (Gastrointestinal disorders) | 15
Dehydration (Metabolism and nutrition disorders) | 2
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 7
Dry mouth (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 3
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 22
Taste disturbance (Nervous system disorders) | 3
Vomiting (Gastrointestinal disorders) | 9
Edema: limb (General disorders) | 6
Alkaline phosphatase increased (Investigations) | 4
AST increased (Investigations) | 8
Bilirubin increased (Investigations) | 2
Creatinine increased (Investigations) | 16
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 2
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Neuropathy-sensory (Nervous system disorders) | 4
Back, pain (Musculoskeletal and connective tissue disorders) | 2
Head/headache (Nervous system disorders) | 3
Joint, pain (Musculoskeletal and connective tissue disorders) | 2
Muscle, pain (Musculoskeletal and connective tissue disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Phlebitis (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No